CLINICAL TRIAL: NCT01147432
Title: A Double Blind, Randomized, Placebo-Controlled, Third-Party Open, Modified Cross-Over Study To Examine The Acute Effect Of PF-04427429 On Capsaicin Flare Response In Healthy Volunteers Using EMLA Cream As Positive Control
Brief Title: Acute Response Capsaicin Flare Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B0141006
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Healthy male volunteers; capsaicin challenge; safety; toleration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-04427429 (Experimental)
  Interventions: Drug: PF-04427429; Other: Capsaicin challenge
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Capsaicin challenge
- EMLA (Active Comparator)
  Interventions: Other: EMLA positive control

INTERVENTIONS:
Drug: PF-04427429 — Single dose IV infusion up to 300mg
  Arms: PF-04427429
Other: Capsaicin challenge — Capsaicin challenge: 110 mg (0.075% capsaicin) to be applied at pre-dose and at 2h, 5h, 8h and 24h post-dose as well as 1 week and 4 weeks post final treatment period
  Arms: PF-04427429
Drug: Placebo — Placebo IV infusion (saline) to be administered during two of the three treatment periods
  Arms: Placebo
Other: Capsaicin challenge — Capsaicin challenge: 110 mg (0.075% capsaicin) to be applied at pre-dose and at 2h, 5h, 8h and 24h post-dose as well as 1 week and 4 weeks post final treatment period
  Arms: Placebo
Other: EMLA positive control — 2g EMLA cream to be applied ONCE during study period 1
  Arms: EMLA

SUMMARY:
Prior to administering PF-04427429 to patients we wish to increase the understanding of functional effects associated with calcitonin gene related peptide (CGRP) pathways. This study will examine whether it is possible for a single dose of PF-04427429 to acutely attenuate a capsaicin induced flare response.

DETAILED DESCRIPTION:
Proof of mechanism in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 50 years inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Skintype I-III with a distance from base of scaphoid to antecubital fossa >26cm on their forearms.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, genitourinary, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, symptomatic, seasonal allergies at time of dosing).
* Use of biologics including any live vaccines within 3 months prior to screening or prior treatment with an antibody in a previous clinical trial or treatment with an immunoglobulin in the past 6 months.
* 12-lead ECG demonstrating QTcF >450 msec at screening.
* Subjects with scars or tattoos on the forearms, or with evidence of sunburn, or excessive hairy volar forearms.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Mean blood perfusion induced by capsaicin challenge, between 30 and 60 minutes post each administration of capsaicin | 7 weeks post first dose

SECONDARY OUTCOMES:
Adverse Events including dose site reactions, blood pressure, pulse rate, ECG, ADA and laboratory safety | 12 weeks post final dose
Plasma concentrations of free PF-04427429 | 6 weekly following week 15
Plasma concentrations of free and total CGRP | 6 weekly following week 15
Mean blood perfusion induced by capsaicin challenge, between 40 and 60 minutes post each administration of capsaicin. | 7 weeks post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0141006&StudyName=Acute%20Response%20Capsaicin%20Flare%20Study%20